CLINICAL TRIAL: NCT00768521
Title: A Randomized, Placebo Controlled, Crossover Study to Evaluate the Effects of Tolterodine Tartrate on Urodynamic Parameters in Patients With Overactive Bladder
Brief Title: A Study to Test the Effects of Tolterodine Tartrate in Patients With Overactive Bladder (0000-107)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-107; 2008_560
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): Part I, Sequence 1: tolterodine tartrate crossing over to matching placebo
  Interventions: Drug: tolterodine tartrate; Drug: Comparator: Placebo to tolterodine tartrate
- 2 (Experimental): Part I, Sequence 2: placebo crossing over to study drug 4 mg once a Day (qd)
  Interventions: Drug: tolterodine tartrate; Drug: Comparator: Placebo to tolterodine tartrate
- 3 (Experimental): Part II, Sequence 1: study drug crossing over to placebo
  Interventions: Drug: tolterodine tartrate; Drug: Comparator: Placebo to tolterodine tartrate
- 4 (Experimental): Part II, Sequence 2: placebo crossing over to study drug
  Interventions: Drug: tolterodine tartrate; Drug: Comparator: Placebo to tolterodine tartrate

INTERVENTIONS:
Drug: tolterodine tartrate — Part I: tolterodine tartrate 4 mg capsule once a day (qd) for 7 days
  Part IIa: tolterodine tartrate 4 mg capsule qd for 7 days
  Part IIb: single dose tolterodine tartrate 4 mg capsule
Drug: Comparator: Placebo to tolterodine tartrate — Part I: placebo to tolterodine tartrate 4 mg capsule once a day (qd) for 7 days
  Part IIa: placebo to tolterodine tartrate 4 mg capsule qd for 7 days
  Part IIb: single dose placebo to tolterodine tartrate 4 mg capsule

SUMMARY:
This study will design an alternative urodynamic platform to better evaluate treatment effects of medications for overactive bladder. Part II is dependent on results of Part I and may not be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a postmenopausal female 40 to 75 years of age
* Patient has a Body Mass Index (BMI) less than or equal to 35 kg/m2
* Patient has a documented history of overactive bladder for at least 6 months prior to screening

Exclusion Criteria:

* Patient has stress or mixed incontinence
* Patient has a history of interstitial cystitis, painful bladder syndrome, or chronic pelvic pain
* Patient has a history of stroke, seizures, or major neurological disorders
* Patient has a history of fecal incontinence
* Patient has a history of continual urine leakage
* Patient has had surgery to correct stress urinary incontinence or pelvic organ prolapse within 6 months of study start
* Patient received bladder training of electrostimulation within 2 weeks of study start
* Patient requires a catheter
* Patient is taking medications that cannot be stopped for the duration of the trial including certain anticholinergics or smooth muscle relaxants
* Patient began taking tricyclic antidepressants, serotonin/norepinephrine reuptake inhibitors, calcium channel blockers, ephedrine/pseudoephedrine, or diuretic therapy less than 8 weeks before study start
* Patient has been on hormone replacement therapy for less than 12 weeks at study start
* Patient must take medication for arrhythmia
* Patient consumes more than 2 alcoholic beverages per day
* Patient consumes more than 3 servings of caffeinated beverages per day (1 serving = 120 mg caffeine)
* Patient has multiple and/or severe allergies to foods and drugs
* Patient regularly uses any illegal drugs

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-09-03 (Actual); Primary Completion 2009-01-19 (Actual); Study Completion 2009-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Frenkl T, Railkar R, Shore N, Bailen J, Sutherland S, Burke J, Scott BB, Ruddy M, Beals C. Evaluation of an experimental urodynamic platform to identify treatment effects: a randomized, placebo-controlled, crossover study in patients with overactive bladder. Neurourol Urodyn. 2012 Jan;31(1):69-74. doi: 10.1002/nau.21094. Epub 2011 Sep 8. PMID 21905086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Entered: 8 Sep 2008
  Last Patient, Last Visit: 19 Jan 2009
  2 sites Since Part I of the study enrolled sufficiently there was no need to modify the study design nor conduct Part II.
Pre-assignment Details: Patients completed a 1-week screening and 1-week placebo run-in period.
  Patients were randomized Visit 3/Day 1. Patients were excluded if they were unable to adequately complete a diary, number of micturitions was ≤ 8, or number of urge incontinence was ≤ 1 on each diary day.
Groups:
- Tolterodine Then Placebo: Tolterodine 4 mg then Placebo
- Placebo Then Tolterodine: Placebo then Tolterodine 4 mg
Period: Period 1
Arm/Group | Tolterodine Then Placebo | Placebo Then Tolterodine
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Tolterodine Then Placebo | Placebo Then Tolterodine
Started | 9 | 11
Completed | 9 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All Study Participants from all groups.
Arm/Group | All Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 59.1 [45 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Maximum Cystometric Capacity at 4 Hours Post Dose 7 on Tolterodine 4 mg and Placebo
Description: Change from baseline in maximum cystometric capacity at 4 hours post dose 7 on tolterodine 4 mg and placebo (analysis on natural log transformed data)
Time Frame: 4 hours post dose 7
Population: All patients
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage change
Groups:
- Tolterodine: Tolterodine 4 mg
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 20 | 20
Percentage change | 1.15 (0.06) [1.04 to 1.28] | 0.94 (0.06) [0.84 to 1.04]
Statistical Analysis 1: Comparison: Tolterodine vs Placebo; Test type: Superiority or Other; p = 0.008, ANCOVA — 1-sided, alpha = 0.05; Baseline used as covariate; Mean Difference (Final Values) = 23.18, 90% CI [7.58 to 41.06] — Primary Hypothesis: Tolterodine LA 4 mg is superior to placebo with respect to change from baseline in maximum cystometric capacity at 4 hours post Dose 7 (i.e., steady state). The expected treatment effect is targeted at 40 mL

2. Secondary Outcome: Change From Baseline in Maximum Cystometric Capacity at 4 Hours Post Dose 1 on Tolterodine 4 mg and Placebo
Description: Change from baseline in maximum cystometric capacity at 4 hours post dose 1 on tolterodine 4 mg and placebo (analysis on natural log transformed data)
Time Frame: 4 hours post dose 1
Population: All patients
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage change
Arm/Group | Tolterodine | Placebo
Number analyzed (Participants) | 20 | 20
Percentage change | 0.92 (0.06) [0.83 to 1.02] | 0.91 (0.06) [0.82 to 1.00]
Statistical Analysis 1: Comparison: Tolterodine vs Placebo; Test type: Superiority or Other; p = 0.422, ANCOVA — 1-sided, alpha = 0.05; Baseline used as covariate; Mean Difference (Final Values) = 1.63, 90% CI [-11.5 to 16.71]

ADVERSE EVENTS:
Time Frame: The adverse experiences reporting are from the randomization visit to follow-up phone call.
Description: Urinalysis and vital sign measurements were performed to monitor safety at clinic visits. Patients were also, queried for any adverse experiences at each visit.
Arm/Group | Tolterodine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolterodine (N=20) | Placebo (N=20)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The analysis presented includes all patients. An analysis excluding patients who were misdosed yielded different results with a similar conclusion and are not presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.